CLINICAL TRIAL: NCT01205971
Title: Oral Health Advocates in Public Housing
Brief Title: Tooth Smart Healthy Start: Oral Health Advocates in Public Housing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Michelle Henshaw, Professor, Boston University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-27749; U54DE019275 (NIH)
Record Dates: First submitted 2010-09-19; First posted 2010-09-21 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Dental Caries in Children
Keywords: Motivational interviewing; Community-based multimodal intervention; Dental Health Advocates; Prevention of ECC; Randomized clinical trial
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing (Experimental): Motivational Interviewing to reduce caregiver risk factors for early childhood caries in their children is delivered by Dental Health Advocates (trained public housing residents) in combination with fluoride varnish applications, oral health assessments and referrals for children.
  Interventions: Behavioral: Motivational Interviewing
- Dental Preventive Services (Active Comparator): Fluoride varnish applications, written oral health educational materials regarding early childhood caries prevention, oral health assessments and referrals.
  Interventions: Behavioral: Dental Preventive Services

INTERVENTIONS:
Behavioral: Motivational Interviewing — Motivational interviewing is delivered by trained public housing residents, every 3 months for a total of 8 sessions over 24 months.
  Arms: Motivational Interviewing
Behavioral: Dental Preventive Services — Written oral health educational materials
  Arms: Dental Preventive Services

SUMMARY:
Dental caries is the most common chronic disease of childhood and is increasing in prevalence in children 2-5 years old. Racial and ethnic minority groups as well as economically disadvantaged individuals are affected the most by this health outcome. This study will test if a community-based multimodal intervention will reduce 2-year incidence of early childhood caries (ECC) in children aged 0-5 living in public housing developments. The intervention combines the components of motivational interviewing (counseling) delivered by dental health advocates, fluoride varnish application, oral health assessment and referral. The investigators hypothesize that the multimodal intervention with motivational interviewing will reduce ECC behavioral risk factors thereby leading to a reduction of ECC incidence when compared to fluoride varnish application, written oral health education materials and oral health assessment and referral.

DETAILED DESCRIPTION:
Dental caries is the most common, chronic disease of childhood, is increasing in prevalence, and disproportionately affects individuals who are financially disadvantaged and from racial and ethnic minority groups. Given the chronic nature of dental caries, clinically based preventive and restorative care alone will likely be inadequate to decrease disparities in early childhood caries (ECC) prevalence. We posit that a multimodal community-based approach, which addresses the chronic, infectious and multifactorial nature of dental caries, will be more effective than either behavioral counseling and the chemotherapeutic effects of fluoride alone. In addition to counseling and fluoride application, a successful community-based multimodal intervention will also need to equip caregivers with the skills to become involved in the prevention and management of ECC.

This group randomized clinical trial will test if a community-based multimodal intervention will reduce the 2-year ECC incidence of children aged 0-5 living in public housing developments. The intervention combines evidence based components and a unique delivery setting (public housing). We hypothesize that the multimodal intervention comprised of oral health assessment and feedback, fluoride varnish application, and motivational interviewing delivered by Dental Health Advocates (trained public housing residents) can reduce incidence of ECC in 0-5 year olds compared with a control group that receives oral health assessment and feedback, fluoride varnish application, and written oral health education materials.

This study is well poised for dissemination. Ultimately, this work could be disseminated nationwide and could potentially improve the oral health of over 500,000 family households and over 1 million children living in public housing.

ELIGIBILITY:
Inclusion Criteria:

* be living in participating public housing sites
* have one or more children 0-5 years old or be in their third trimester of pregnancy
* plan to live in their current housing development for the ensuing 24 months
* be able and willing to provide informed consent

Exclusion Criteria:

* caregivers unable to communicate orally in English or Spanish
* subject child has a known systemic disease associated with abnormal tooth development or abnormal oral health status such as cleft lip or palate, Burkett's lymphoma, osteogenesis imperfecta, ameliogenesis imperfecta, or dentinogenesis imperfecta
* children who have a known allergy to fluoride varnish and its components
* caregivers less than 15 years old

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2842 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2016-12-23 (Actual); Study Completion 2016-12-23 (Actual)

PRIMARY OUTCOMES:
Dental caries incidence | 24 months

SECONDARY OUTCOMES:
Behavioral risk factors for early childhood caries | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Michelle M Henshaw, DDS, MPH, Principal Investigator — Boston University; Belinda Borrelli, PhD, Principal Investigator — Brown University
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers can make a data request through the EC4 website oralhealthdisparities.ucsf.edu

REFERENCES:
- [Derived] Henshaw MM, Borrelli B, Gregorich SE, Heaton B, Tooley EM, Santo W, Cheng NF, Rasmussen M, Helman S, Shain S, Garcia RI. Randomized Trial of Motivational Interviewing to Prevent Early Childhood Caries in Public Housing. JDR Clin Trans Res. 2018 Oct;3(4):353-365. doi: 10.1177/2380084418794377. Epub 2018 Aug 22. PMID 30238060
- [Derived] Albino J, Tiwari T, Gansky SA, Henshaw MM, Barker JC, Brega AG, Gregorich SE, Heaton B, Batliner TS, Borrelli B, Geltman P, Kressin NR, Weintraub JA, Finlayson TL, Garcia RI; Early Childhood Caries Collaborating Centers. The basic research factors questionnaire for studying early childhood caries. BMC Oral Health. 2017 May 19;17(1):83. doi: 10.1186/s12903-017-0374-5. PMID 28526003
- See also: Northeast Center for Research to Evaluate and Eliminate Dental Disparities — http://www.bu.edu/creedd